CLINICAL TRIAL: NCT02213484
Title: Micro RNAs as a Marker of Aortic Aneurysm in Hereditary Aortopathy Syndromes
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0567; UL1TR001082 (NIH)
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Marfan Syndrome; Loeys-Dietz Syndrome; Thoracic Aortic Aneurysm and Dissection Syndromes; Ehlers-Danlos Type IV Syndrome; Turner Syndrome
Keywords: aortopathy syndrome; aortic aneurysm; aortic dissection; connective tissue disorder
MeSH Terms: conditions — Marfan Syndrome; Loeys-Dietz Syndrome; Aortic Aneurysm, Thoracic; Ehlers-Danlos Syndrome, Type IV; Turner Syndrome; Aortic Aneurysm; Aortic Dissection; Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fractionated blood samples will be retained at a part of the study including plasma, platelets and mononuclear cells. At this time genetic testing (genotyping) of individual biospecimens is not included in the IRB-approved protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Marfan syndrome: Individuals with a clinical diagnosis of Marfan syndrome
- Aortopathy syndrome: Individuals with one of the following clinical diagnoses: Loeys-Dietz syndrome, Turner syndrome, Ehlers-Danlos type IV syndrome, Thoracic Aortic Aneurysm and Dissection syndromes.

SUMMARY:
The primary objective of this study is to determine whether specific patterns of circulating micro-ribonucleic acids (miRNAs) are associated with aortic aneurysm and dissection in patients with hereditary aortopathy syndromes. The most common of these syndromes is Marfan Syndrome (MFS), but several other recognized aortopathy syndromes are well characterized. The investigators propose the use of a simple blood test, from which miRNA profiles can be measured in individuals with aortopathy syndromes to be compared with miRNAs observed in a control population that has no known predisposition for aortic disease. The investigators hypothesize that microRNA profiles in individuals with Marfan syndrome, and related disorders, will be distinct from those seen in a control group. The investigators predict that up- or down-regulation of certain miRNAs will correlate with the presence and severity of aortic aneurysm, responses to medical therapy, and ultimately could be used to determine when an individual may be at risk of dissection.

ELIGIBILITY:
Inclusion Criteria: To be in the study, the participant must meet the following criteria

1. Diagnosis of hereditary aortopathy based upon:

   * Confirmation of a disease causing mutation in a known aortopathy disorder OR
   * Confirmation of disease based on published clinical criteria
2. Participants is male or female and greater than 30 days old
3. Participants are able to undergo standard of care cardiac monitoring including an echocardiogram
4. Willing and able to provide written informed consent by parent(s) or guardian(s) after the nature of the study has been explained and prior to any research related procedures
5. Signed HIPPA compliant research authorization

Exclusion Criteria: Participant will be excluded from the study for any of the following criteria

1. Diagnosis of a hereditary aortopathy can not be confirmed
2. Existence of an additional comorbid condition- including a co-existing genetic syndrome, heart failure, renal disease, rheumatologic disease, history of malignancy, thyroid disease, recent stroke, other life-limiting illness not related to cardiovascular disease.
3. Extreme prematurity, <28 weeks gestational age

Ages: 30 Days to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All individuals up to 60 years seen in the Children's Hospital of Colorado and University Hospital Marfan Syndrome Clinics will be eligible for enrollment in this study. Individuals with a clinical diagnosis of Marfan syndrome with or without genetic confirmation will be included as will patients with recognized aortopathy syndromes or family history of aortopathy with evidence of aorta disease. Subjects will be primarily recruited through the Heart Institute at Children's Hospital Colorado and through the cardiology team at the University of Colorado Hospital. Pediatric patients with Marfan syndrome and related aortopathy syndromes are primarily followed in the Principal Investigator, Dr. Chatfield's, Cardiac Genetics Clinic at Children's Hospital Colorado and will be recruited from this clinic. Adult patients with aortopathy syndromes are followed primarily in the Adult Congenital Heart Disease Clinic at University of Colorado Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Plasma miRNA profiling in individuals with Marfan syndrome | 2 years
  In a cross-sectional analysis, characterize circulating miRNA profiles in individuals with Marfan syndrome and compare to profiles in normal age-matched controls.
Plasma miRNA profiling in individuals with aortopathy syndromes | 3 years
  In a cross-sectional analysis, characterize circulating miRNA profiles in individuals with aortopathy syndromes and compare to profiles in normal age-matched controls.

SECONDARY OUTCOMES:
Correlation of plasma miRNA profiles with aortic dimensions | 2 years
  In a cross-sectional analysis correlate miRNA profiles with aortic dimension and Z-score, type of medication used, history of aneurysm and/or dissection, and need for surgical intervention in individuals with MFS.

OTHER OUTCOMES:
Correlation of plasma miRNA with progression of aortic aneurysm | 5 years
  Correlate miRNA patterns with changes in aortic dimension and Z-score longitudinally at yearly time points.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn C Chatfield, MD, PhD, Principal Investigator — University of Colorado Denver, Children's Hospital Colorado
Locations (2):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado